CLINICAL TRIAL: NCT04466332
Title: Comparison of Two ECG Guided PICC Insertion Techniques, a Randomized Controlled Trial
Brief Title: Comparison of Two ECG Guided PICC Insertion Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Salah D. Qanadli, MD, PhD, Professor MD PhD, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-00583
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Central Venous Access; Long Term Antibiotics; Chemotherapy; Total Parenteral Nutrition
Keywords: PICC; ECG guidance; Central Venous Catheter; Catheterization
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline ECG with Pilot Tip Location System (Experimental): PICC insertion using electrocardiographic guidance Pilot Tip Location System (TLS), ECG signal transmission is with saline water
  Interventions: Device: LifeCath-CT PICC easy™ (Vygon)
- Guidewire ECG with Sherlock Tip Confirmation System (Experimental): PICC insertion using electrocardiographic guidance Sherlock 3CG Tip Confirmation System (TCS), ECG signal transmission is with guidewire
  Interventions: Device: PowerPICC-SOLO® (C.R. Bard)

INTERVENTIONS:
Device: LifeCath-CT PICC easy™ (Vygon) — ECG electrodes are placed on patient's chest ensuring that there is a distinguishable P-wave.
  Upper arm selection is based on vein diameter and dominance, ultrasound is used to identify a suitable vein.
  The patient is prepared using a maximal sterile barrier approach. The catheter is inserted into one of the veins (75-90° arm abduction) using ultrasound and modified Seldinger technique.
  The PICC is advanced into the central circulation and used as an intracavitary electrode (connection with Vygocard2™). Saline water instilled through the catheter ensures conductivity.
  The ECG is then used until displayed intracavitary P-wave has a maximal height without negative deflexion. Catheter is left at this point (cavo atrial junction).
  The PICC hub side is then trimmed and the catheter part connected. The PICC is caped with a neutral bidirectional valve.
  The puncture site is dressed and catheter stabilized. Chest Xray is obtained immediately after insertion to assess the position.
  Arms: Saline ECG with Pilot Tip Location System
Device: PowerPICC-SOLO® (C.R. Bard) — ECG electrodes are placed on patients chest ensuring that there is a distinguishable P-wave.
  Upper arm selection is based on vein diameter and dominance, ultrasound is used to identify suitable vein.
  The patient is prepared using a maximal sterile barrier approach. The catheter is inserted into one of the veins (75-90° arm abduction) using ultrasound and modified Seldinger technique.
  The catheter's free end is cut to the anticipated length using anthropometric measurements (insertion/axillary crease+axillary crease/sternal notch+13cm) and the preloaded magnetic-tipped stylet (serving as intracavitary electrode) is put inside.
  The PICC is advanced into central veins until intravascular ECG displays a P-wave with maximal height without negative deflexion. Catheter is left at this point (cavo atrial junction).
  The puncture site is dressed and catheter stabilized. Chest Xray is obtained immediately after insertion to assess position.
  Arms: Guidewire ECG with Sherlock Tip Confirmation System

SUMMARY:
The aim of our study is to compare two ECG techniques for guiding Peripherally Inserted Central Venous Cather (PICC) in terms of accuracy of the final position of the catheter tip.

DETAILED DESCRIPTION:
One technique uses ECG signal transmission with saline water and allows external catheter length adjustment while the other technique uses a guidewire for signal transmission thus requiring prior catheter length adjustment

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Adult > 18 years
* Referred to the interventional radiology department for PICC insertion

Exclusion Criteria:

* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Impairment of the heart rhythm changing the presentation of the P wave (atrial fibrillation, atrial flutter, severe tachycardia, pacemaker driven rhythm)
* Enrolled in conflicting research study
* Weight> 150 kg, technical limit for the fluoroscopy table
* Impossibility of obtaining informed consent
* Refusal to be informed in the event of a chance discovery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Distance from catheter tip to cavo-atrial junction (CAJ) | At the end of intervention
  At the end of intervention tip position is measured on chest fluoroscopic X-ray.
  Absolute distance in centimeters from tip to CAJ is measured on the image

SECONDARY OUTCOMES:
Length of the outgoing catheter | At the end of intervention
  Length of the outgoing catheter at the entry point near the bend of the elbow in centimeters
Haemostasis time | At the end of intervention
  Haemostasis time at the puncture site entry point (0, 1, 3, 5, >5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Salah Dine Qanadli, Prof. MD PhD, Study Director — UNIL-CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No